CLINICAL TRIAL: NCT03302988
Title: Wound Eversion Versus Planar Closure for Wounds on the Face or Neck: a Randomized Split Wound Comparative Effectiveness Trial
Brief Title: Wound Eversion Versus Planar Closure for Face or Neck Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 803389
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Operative Wound
Keywords: Wound Edge Eversion; Dermal Sutures
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Each wound will have 2 treatments. The type of treatment (Type of suturing) will be chosen by random assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Everted closure (Experimental): Wound eversion will be achieved through buried vertical mattress suture or cuticular suture based on surgeon's preference, either buried vertical mattress suture or cuticular sutures
  Interventions: Other: Everted closure
- Planar closure (Active Comparator): The planar side of the same wond will be closed with traditional buried simple closure and running cuticular sutures
  Interventions: Other: Planar closure

INTERVENTIONS:
Other: Everted closure — Suturing technique to obtain wound eversion. Type of suturing technique at surgeon's discretion
  Arms: Everted closure
Other: Planar closure — The planar side will be closed with traditional buried simple closure and running cuticular sutures
  Arms: Planar closure

SUMMARY:
The aim of this study is to determine whether wound edge eversion, achieved by careful placement of dermal sutures, improves the cosmetic outcome of operative wounds closed on the head or neck.

DETAILED DESCRIPTION:
It has been established that as wounds heal, the resultant tissue remodeling results in wound contracture. Surgeons are taught that by everting wounds' edges with well-placed dermal sutures, there is less depression of the resultant scar. A prior study conducted by us at this center found that wound eversion was not associated with better cosmetic outcome (1). However, it was noted that most of the procedures were performed off the head and neck, places where the effects of eversion were thought to be most beneficial (2) Thus our goal is to now study the effects of eversion exclusively on the face and neck.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure with predicted linear closure on the face or neck
* Willing to return for follow up visits

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Patient Observer Scar Assessment Scale (POSAS) | Within 3 months
  The primary endpoint will be the score of two blinded reviewers using the physician observer assessment score at a three-month assessment visit.
Incidence of sunken scars | Within 3 months
  The incidence of sunken scars or elevated scaring on each treatment side will also be determined

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kappel S, Kleinerman R, King TH, Sivamani R, Taylor S, Nguyen U, Eisen DB. Does wound eversion improve cosmetic outcome?: Results of a randomized, split-scar, comparative trial. J Am Acad Dermatol. 2015 Apr;72(4):668-73. doi: 10.1016/j.jaad.2014.11.032. Epub 2015 Jan 23. PMID 25619206
- [Background] Trufant JW, Leach BC. Commentary: Wound edge eversion: surgical dogma or diversion? J Am Acad Dermatol. 2015 Apr;72(4):681-2. doi: 10.1016/j.jaad.2014.09.046. No abstract available. PMID 25773410
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683